CLINICAL TRIAL: NCT01042509
Title: Combination of Alemtuzumab (Anti-CD52) and Rituximab (Anti-CD20) at Low-doses in Chronic Graft Versus Host Disease Treatment After First-line Therapy Failure.
Brief Title: Combination of Alemtuzumab and Rituximab at Low-doses in Refractory Chronic Graft-Versus-Host Disease
Acronym: LowAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, Dr., Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE09-013
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-12

CONDITIONS: Graft vs Host Disease
Keywords: Chronic Graft vs Host Disease; Alemtuzumab; Rituximab; Low-dose; Alemtuzumab and rituximab combination
MeSH Terms: conditions — Graft vs Host Disease | interventions — Alemtuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alemtuzumab and rituximab (Experimental): Patients with chronic GVHD after first-line therapy failure will receive Alemtuzumab at 10mg subcutaneously daily for 3 doses (days 1, 2 and 3) Rituximab at 100mg intravenously weekly for 4 doses (days 4, 11, 18 and 25. THE STUDY HAVE ONLY ONE ARM.
  Interventions: Drug: Alemtuzumab and rituximab

INTERVENTIONS:
Drug: Alemtuzumab and rituximab — Alemtuzumab at 10mg subcutaneously daily for 3 doses (days 1, 2 and 3) Rituximab at 100mg intravenously weekly for 4 doses (days 4, 11, 18 and 25
  Other Names: Campath; Rituxan

SUMMARY:
The purpose of this study is to determine whether low-doses alemtuzumab and rituximab combination are effective in the treatment of chronic graft-versus-host disease (GVHD) after first-line therapy failure.

DETAILED DESCRIPTION:
Graft-versus-host disease (GVHD) is the most common long-term complication in patients who underwent allogeneic transplantation. First-line therapy for chronic GVHD is based on immunosuppressive agents (usually cyclosporine and corticosteroids) achieving satisfactory response in around 30% of patients. There is no ideal second-line treatment for chronic GVHD; however, numerous studies have been published with therapeutic options such as alemtuzumab (anti-CD52) and rituximab (anti-CD20).

This is a prospective, longitudinal, nonrandomized study in which alemtuzumab and rituximab will be administered at low-doses to patients with refractory chronic GVHD. Clinical response will be evaluated based on the Working Group Report 2006, published by the National Institute of Health Consensus. Follow-up sessions will be weekly for four weeks, every two weeks until achieve response, and finally every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic graft-versus-host disease.
* Patients over 18 years old.
* Patients who received first-line treatment with no response (failure), relapse or steroid dependance.

Exclusion Criteria:

* Patients with active bacterial or viral infections.
* Patients with hematologic disease progression.
* Patient's intolerance to drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez-Almaguer, M.D., Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hematology Department of Hospital Universitario Dr Jose E Gonzalez, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Pavletic SZ, Martin P, Lee SJ, Mitchell S, Jacobsohn D, Cowen EW, Turner ML, Akpek G, Gilman A, McDonald G, Schubert M, Berger A, Bross P, Chien JW, Couriel D, Dunn JP, Fall-Dickson J, Farrell A, Flowers ME, Greinix H, Hirschfeld S, Gerber L, Kim S, Knobler R, Lachenbruch PA, Miller FW, Mittleman B, Papadopoulos E, Parsons SK, Przepiorka D, Robinson M, Ward M, Reeve B, Rider LG, Shulman H, Schultz KR, Weisdorf D, Vogelsang GB; Response Criteria Working Group. Measuring therapeutic response in chronic graft-versus-host disease: National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. Response Criteria Working Group report. Biol Blood Marrow Transplant. 2006 Mar;12(3):252-66. doi: 10.1016/j.bbmt.2006.01.008. PMID 16503494
- [Background] Martin PJ, Weisdorf D, Przepiorka D, Hirschfeld S, Farrell A, Rizzo JD, Foley R, Socie G, Carter S, Couriel D, Schultz KR, Flowers ME, Filipovich AH, Saliba R, Vogelsang GB, Pavletic SZ, Lee SJ; Design of Clinical Trials Working Group. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: VI. Design of Clinical Trials Working Group report. Biol Blood Marrow Transplant. 2006 May;12(5):491-505. doi: 10.1016/j.bbmt.2006.03.004. PMID 16635784
- [Background] Ruiz-Arguelles GJ, Gil-Beristain J, Magana M, Ruiz-Delgado GJ. Alemtuzumab-induced resolution of refractory cutaneous chronic graft-versus-host disease. Biol Blood Marrow Transplant. 2008 Jan;14(1):7-9. doi: 10.1016/j.bbmt.2007.09.013. Epub 2007 Dec 3. PMID 18158955
- [Background] Zaja F, Bacigalupo A, Patriarca F, Stanzani M, Van Lint MT, Fili C, Scime R, Milone G, Falda M, Vener C, Laszlo D, Alessandrino PE, Narni F, Sica S, Olivieri A, Sperotto A, Bosi A, Bonifazi F, Fanin R; GITMO (Gruppo Italiano Trapianto Midollo Osseo). Treatment of refractory chronic GVHD with rituximab: a GITMO study. Bone Marrow Transplant. 2007 Aug;40(3):273-7. doi: 10.1038/sj.bmt.1705725. Epub 2007 Jun 4. PMID 17549053
- [Background] von Bonin M, Oelschlagel U, Radke J, Stewart M, Ehninger G, Bornhauser M, Platzbecker U. Treatment of chronic steroid-refractory graft-versus-host disease with low-dose rituximab. Transplantation. 2008 Sep 27;86(6):875-9. doi: 10.1097/TP.0b013e318183f662. PMID 18813113
- [Derived] Gutierrez-Aguirre CH, Cantu-Rodriguez OG, Borjas-Almaguer OD, Gonzalez-Llano O, Jaime-Perez JC, Solano-Genesta M, Gomez-Guijosa M, Mancias-Guerra C, Tarin L, Gomez-Almaguer D. Effectiveness of subcutaneous low-dose alemtuzumab and rituximab combination therapy for steroid-resistant chronic graft-versus-host disease. Haematologica. 2012 May;97(5):717-22. doi: 10.3324/haematol.2011.054577. Epub 2011 Dec 1. PMID 22133770

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Chronic GVHD: Patients with chronic GVHD after first-line therapy failure.
Period: Overall Study
Arm/Group | Patients With Chronic GVHD
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Chronic GVHD
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (20)
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  Mexico | 15

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response of Patients With Refractory Chronic GVHD Based on the Working Group Report 2006.
Description: Overall response of participants to alemtuzumab and rituximab combination at day +30, +90 and +365 of follow-up
Time Frame: 30, 90 and 365 days
Population: All consecutive patients were included in an intention to treat analysis to evaluate clinical response to alemtuzumab and rituximab combination.
Measure: Number; unit: percentage of participants
Groups:
- Treatment Group: This study had only one arm
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
percentage of participants
  Overall response at +30-day evaluation | 100
  Overall response at +90-day evaluation | 78
  Overall response at +365-day evaluation | 80

2. Secondary Outcome: Side Effects
Description: Percentage of participants who experienced side effects
Time Frame: 365 days
Population: 15 consecutive patients were included for the analysis with periodical clinical evaluations to assess adverse effects.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 15
Participants | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 10/15
Other Adverse Events (participants affected / at risk) | 7/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=15)
pneumonia (Infections and infestations) | 1 (1) — pneumonia by Rhodococcus equi
infection (Infections and infestations) | 9 (9) — laryngitis, sinusitis, pneumonia, urinary tract infection and oral herpes simplex virus infection in 1 patient each, bronchitis in 2 and reactivation of cytomegalovirus in 3 patients
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=15)
pneumonia (Investigations) | 7 (7) — Chills, rash an fever

LIMITATIONS AND CAVEATS:
A limitation of this trial is the small number of subjects included

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No